CLINICAL TRIAL: NCT05905159
Title: Neural Mechanisms Underlying Attentional Bias Modification in Fibromyalgia Patients: a Double-blind ERP Study
Brief Title: Attentional Bias Modification in Fibromyalgia Patients (ABM)
Acronym: ABM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ABM-URJC
Record Dates: First submitted 2023-05-30; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Fibromyalgia
Keywords: Attentional bias modification; Dot-Probe Task; Fibromyalgia; ERPs; Pain-related Faces
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABM (Experimental): ABM training will consist of five sessions over five consecutive days during which patients performed a modified version of the visual dot-probe task. The whole ABM program will include a total of 1000 trials that will be distributed in 200 trials per session (twenty minutes per session).
  Participants assigned to ABM training condition will be trained implicitly to attend away from pain-related stimuli (i.e., facial expressions). They will be presented with a modified dot-probe task with trials including targets that often replaced neutral faces. Thus, 80% of trials (i.e., 160 trials) included targets that replaced neutral cue faces (pain incongruent trials: target appeared in the opposite side of pain-related faces). The rest of trials (i.e., 40 trials) belonged to pain congruent trials (i.e., target will occur in the same location of the pain-related facial expression).
  Interventions: Behavioral: ABM
- Control (Placebo Comparator): By contrast, patients assigned to control condition were exposed to a standard visual dot-probe task in which targets were equally likely to replace pain or neutral cues (i.e., facial expressions) during pain trials (i.e., 50% pain-incongruent trials and 50% pain-congruent tri-als). The whole Control program will include a total of 1000 trials that will be distributed in 200 trials per session (twenty minutes per session).
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: ABM — Direct attention away from pain-related information (i.e., facial expressions) through implicit training procedures
  Arms: ABM
Behavioral: Control — Direct attention equally towards pain-related and neutral information (i.e., facial expressions) through implicit training procedures
  Arms: Control

SUMMARY:
There is a growing interest in the potential benefits of attentional bias modification (ABM) training in chronic pain patients. However, studies examining the effectiveness of ABM programs in fibromyalgia patients have demonstrated inconclusive effects on both behavioral indices and clinical symptoms. Underlying neural dynamics of ABM effects could yield additional insights but remain yet unexplored.

Current study, therefore, aimed investigating the effects of ABM training on known neural indicators of attentional bias to pain using electroencephalography (EEG).

The goal of this clinical trial is to test the effects of ABM training on known neural indicators of attentional bias to pain using electroencephalography (EEG) in fibromyalgia patients

The main question[s] it aims to answer are:

* Are fibromyalgia patients sensitive to ABM procedures?
* What are the neural indices associated with ABM procedures?
* Do ABM procedures transfer of effects on the clinical symptomatology in fibromyalgia patients?

Participants will performes five sessions consisting of a modified dot-probe task in which patients were trained to avoid facial pain expressions, whereas in the control group participants will performes five sessions consisting of a standard dot-probe task. Potential ABM training effects will be evaluated by comparing a single pre- and post-treatment session, in which event-related potentials (ERPs) will be recorded in response to three experimental tasks (standard dot-probe, RIR, and visual tasks).

Furthermore, patients will fill a series of self-report questionnaires assessing anxiety, depression, pain-related worrying, fear of pain, fatigue and pain status.

Researchers will compare two fibromyalgia patients groups that will enrolled and randomly assigned to an ABM training in order to see attentional improvements in the training fibromyalgia group.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia Diagnosis.
* Female sex
* The presence of clinical symptoms regarding anxiety or depression will be not exclusion criteria, as long as fibromyalgia was participants' primary diagnosis.

Exclusion Criteria:

* Participation in the study will require the absence of neurological and psychiatric disorders that impair cognitive functions (i.e., stroke brain damage, psychosis, bipolar disorder, and substance abuse/dependence).
* Pregnancy
* Not being able to read Spanish in order to fill in the questionnaires

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Attentional bias from baseline (pre-training) | Behavioural Attentional bias from baseline (pre-training)
  Attentional bias will be assessed by dot-probe task. Behavioural reaction times outcomes will be recorder. The reaction time average for each dot-probe condition will be included as intrasubject factor and the training group as between-subject factor.
Attentional bias from baseline (pre-training) | ERPs Attentional bias from baseline (pre-training)
  Attentional bias will be assessed by dot-probe task. Event-related potentials (ERPs) outcomes will be recorder. The P2 and N2 ERPs average amplitudes for each dot-probe condition will be included as intrasubject factor and the training group as between-subject factor.
Changes on Attentional bias from baseline (pre-training) to 1 day post-training | Behavioural attentional bias modification changes from baseline (pre-training vs 1 day post-training)
  Attentional bias will be assessed by dot-probe task. Behavioural reaction times outcomes will be recorder. To test the effect of the ABM procedure, the reaction time average for each dot-probe condition will be included as intrasubject factor and the training group as between-subject factor.
Changes on Attentional bias from baseline (pre-training) to 1 day post-training | ERPs attentional bias modification changes from baseline (pre-training vs 1 day post-training)
  Attentional bias will be assessed by dot-probe task. ERPs outcomes will be recorder. To test the effect of the ABM procedure, ERPs amplitudes for each dot-probe condition will be included as intrasubject factor and the training group as between-subject factor.

SECONDARY OUTCOMES:
Anxiety scores from baseline (pre-training) to 1 day post-training | Anxiety scores from baseline changes from baseline (pre-training vs 1 day post-training)
  Anxiety will be assessed by the Spanish version of the State-Trait Anxiety Inventory (STAI) questionnaire. The scale include 20 items and are scored using a four-point Likert scale, ranging from 0 to 3. Higher scores (i.e., > 60 percentile) represents high anxiety levels. Anxiety scores will be included as intrasubject factor and the training group as between-subject factor.
Depression scores from baseline (pre-training) to 1 day post-training | Depression scores from baseline changes from baseline (pre-training vs 1 day post-training)
  Depression will be assessed by the Spanish version of the Beck Depression Inventory (BDI). The scale include 21 items with four different statements describing various degrees of symptom intensity. Higher scores (i.e., > 21) represents greater severity of depressive symptoms. Depression scores will be included as intrasubject factor and the training group as between-subject factor.
Fear of pain scores from baseline (pre-training) to 1 day post-training | Fear of pain scores from baseline changes from baseline (pre-training vs 1 day post-training)
  Fear of pain will be assessed by the Spanish version of Fear of Pain Questionnaire (FPQ). In FPQ questionnaire participants are asked to rate in 30 items how fearful to pain experiences on a 5-point Likert scale. Higher scores represents greater severity of fear of pain symptoms. Fear of pain scores will be included as intrasubject factor and the training group as between-subject factor.
Pain worrying scores from baseline (pre-training) to 1 day post-training | Pain worrying scores from baseline changes from baseline (pre-training vs 1 day post-training)
  Pain worrying will be assessed by the Spanish versions of the Pain Catastrophizing Scale (PCS). In this scale, participants rated in 13 items the frequency of experiencing each catastrophic belief on a 0 to 4 Likert scale. Higher scores represents greater severity of pain worrying symptoms. Pain worrying scores will be included as intrasubject factor and the training group as between-subject factor.
Fibromyalgia impact scores from baseline (pre-training) to 1 day post-training | Fibromyalgia impact scores from baseline changes from baseline (pre-training vs 1 day post-training)
  Fibromyalgia impact will be assessed by the Spanish version of the Fibromyalgia Impact Questionnaire (FIQ). FIQ consists of 10 items for the assessment of three fibromyalgia domains (function, overall impact and symptoms). Higher scores represents greater severity of fibromyalgia impact symptoms. Fibromyalgia impact scores will be included as intrasubject factor and the training group as between-subject factor.
Pain scores from baseline (pre-training) to 1 day post-training | Pain scores from baseline changes from baseline (pre-training vs 1 day post-training)
  Pain status will be assessed by a visual analogue scale (VAS). The scale include 0 to 10 likert scale. Higher scores (i.e., > 6) represents greater severity of pain intensity symptoms. Pain scores will be included as intrasubject factor and the training group as between-subject factor.
Fatigue scores from baseline (pre-training) to 1 day post-training | Fatigue scores from baseline changes from baseline (pre-training vs 1 day post-training)
  Fatigue status will be assessed by a visual analogue scale (VAS). The scale include 0 to 10 likert scale. Higher scores (i.e., > 6) represents greater severity of fatigue intensity symptoms. Fatigue scores will be included as intrasubject factor and the training group as between-subject factor.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Mercado, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlson JM. A systematic review of event-related potentials as outcome measures of attention bias modification. Psychophysiology. 2021 Jun;58(6):e13801. doi: 10.1111/psyp.13801. Epub 2021 Mar 8. PMID 33682161
- [Background] Eldar S, Bar-Haim Y. Neural plasticity in response to attention training in anxiety. Psychol Med. 2010 Apr;40(4):667-77. doi: 10.1017/S0033291709990766. Epub 2009 Jul 23. PMID 19627649
- [Background] Carleton RN, Asmundson GJG, Korol SL, LeBouthillier DM, Hozempa K, Katz JD, Vlaeyen JWS, Crombez G. Evaluating the efficacy of an attention modification program for patients with fibromyalgia: a randomized controlled trial. Pain. 2020 Mar;161(3):584-594. doi: 10.1097/j.pain.0000000000001746. PMID 31693540
- [Background] Crombez G, Van Ryckeghem DML, Eccleston C, Van Damme S. Attentional bias to pain-related information: a meta-analysis. Pain. 2013 Apr;154(4):497-510. doi: 10.1016/j.pain.2012.11.013. Epub 2012 Dec 5. PMID 23333054
- [Background] Fernandes-Magalhaes R, Ferrera D, Pelaez I, Martin-Buro MC, Carpio A, De Lahoz ME, Barjola P, Mercado F. Neural correlates of the attentional bias towards pain-related faces in fibromyalgia patients: An ERP study using a dot-probe task. Neuropsychologia. 2022 Feb 10;166:108141. doi: 10.1016/j.neuropsychologia.2021.108141. Epub 2022 Jan 4. PMID 34995568
- [Background] Mogoase C, David D, Koster EH. Clinical efficacy of attentional bias modification procedures: an updated meta-analysis. J Clin Psychol. 2014 Dec;70(12):1133-57. doi: 10.1002/jclp.22081. Epub 2014 Mar 20. PMID 24652823
- [Background] Todd J, Sharpe L, Johnson A, Nicholson Perry K, Colagiuri B, Dear BF. Towards a new model of attentional biases in the development, maintenance, and management of pain. Pain. 2015 Sep;156(9):1589-1600. doi: 10.1097/j.pain.0000000000000214. PMID 26291997
- [Derived] Fernandes-Magalhaes R, Carpio A, Ferrera D, Pelaez I, De Lahoz ME, Van Ryckeghem D, Van Damme S, Mercado F. Neural mechanisms underlying attentional bias modification in fibromyalgia patients: a double-blind ERP study. Eur Arch Psychiatry Clin Neurosci. 2024 Aug;274(5):1197-1213. doi: 10.1007/s00406-023-01709-4. Epub 2023 Nov 19. PMID 37980687